CLINICAL TRIAL: NCT05441995
Title: Cryotherapy Efficacy in 9 to17-year-old Children During Endodontic Treatment of the Mandibular First Permanent Molars With Symptomatic Irreversible Pulpitis: a Randomized Parallel Controlled Trial
Brief Title: Cryotherapy Efficacy During Pulp Therapy of the Mandibular First Permanent Molars in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Ahmad Elheeny, Assistant Professor, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 630
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Cryotherapy Effect; Irreversible Pulpitis; Pain
MeSH Terms: conditions — Pain | interventions — Cryotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryotherapy (Experimental)
  Interventions: Other: Cryotherapy
- Inferior alveolar nerve block (Active Comparator)
  Interventions: Other: Cryotherapy

INTERVENTIONS:
Other: Cryotherapy — Ice packs were applied in the buccal mucosa related to the tooth for 5 minutes after IANB administration

SUMMARY:
The aim of the study is to assess the efficacy of cryotherapy application on the success of inferior alveolar nerve block (IANB) in reducing pain during pulp therapy of the mandibular first permanent molars with irreversible pulpitis (IP) in children age from 7 to 16 years. The null hypothesis (H0) supposed no difference in pain intensity during pulp therapy of primary molars with IP anesthetized with IANB with and without cryotherapy application. The secondary aim was to evaluate the children's behavior before and after pulpectomy in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 9-17 years who were categorized as class I or II according to the ASA classification.
* Cooperative children (rate 3 or 4 according to Frankl behavior rating scale)
* Presence of a vital mandibular first permanent molar with SIP, the tooth should show deep caries or dental restorations with a history of spontaneous lingered pain precipitated by thermal stimuli. To confirm the diagnosis of irreversible pulpitis, early response to electric pulp and thermal testing was performed.
* No radiographic changes with at least two-thirds of the root must be evident.

Exclusion Criteria:

* Children with severe emotional, intellectual, and behavioral difficulties.
* Necrotic pulp of primary molars.
* Unrestorable crowns
* Positive history of gingival swelling, abnormal mobility, and fistulous tract.
* Presence of radiographic signs of periapical and/or furcation radiolucency, and pathological resorption.

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | up to 24 hours
  Pain was assessed using Visual Analogue Scale (VAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Minia University, Minya, Minya Governorate, Egypt